CLINICAL TRIAL: NCT03099148
Title: Relative Bioavailability and the Effect of Food on the Bioavailability of LY3337641 in Healthy Subjects
Brief Title: A Study of LY3337641 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16298; I8K-MC-JPDF (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-03-30; First posted 2017-04-04 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3337641 (R-fasted) (Experimental): A single, PO dose of reference formulation (R) given orally with water after an overnight fast in one of four periods.
  Interventions: Drug: Reference Formulation (R)
- LY3337641 (T1-fasted) (Experimental): A single, PO dose of LY3337641(20mg) test formulation 1 (T1) given orally with water after an overnight fast in one of four periods.
  Interventions: Drug: LY3337641 (T1)
- LY3337641 (T1-fed) (Experimental): A single, PO dose of LY3337641 (20mg) test formulation 1 (T1) given orally with water after a high fat meal in one of four periods.
  Interventions: Drug: LY3337641 (T1)
- LY3337641 (T2-fasted) (Experimental): A single, PO dose of LY3337641 (20 mg) test formulation 2 (T2) given orally with water after an overnight fast in one of four periods.
  Interventions: Drug: LY3337641 (T2)

INTERVENTIONS:
Drug: Reference Formulation (R) — Administered PO
  Arms: LY3337641 (R-fasted)
Drug: LY3337641 (T1) — 20 mg PO
  Arms: LY3337641 (T1-fasted); LY3337641 (T1-fed)
Drug: LY3337641 (T2) — 20 mg PO
  Arms: LY3337641 (T2-fasted)

SUMMARY:
The purposes of this study are to determine:

* If there are any differences in the amount of LY3337641 in the blood/body when it is taken in different formulations. A total of 3 different formulations of LY3337641 are being tested.
* How a high-fat meal affects the amount of LY3337641 in the blood/body.
* How safe and well tolerated LY3337641 is.

The study has four periods. Individuals will participate in all four periods. Each period will include 4 overnight stays (5 days) in the Clinical Research Unit (CRU).

This study is expected to last up to 8 weeks. This includes the initial screening period, the study or dosing period, and the follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 18.5 to 32 kilograms per meter squared (kg/m²) inclusive
* Have clinical laboratory test results within normal reference range for the population or investigative site
* Are able and willing to give signed informed consent

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have significant history of or current cardiovascular, dermatological (such as eczema, psoriasis, and acne), respiratory, hepatic, renal, gastrointestinal (cholecystectomy is not acceptable), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have used or intend to use over-the-counter or prescription medication, including herbal medications, within 14 days prior to planned dosing
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Singapore (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Singapore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 period, 4 sequence, randomized crossover study with at least 5 days between doses.
Groups:
- Sequence ADBC: A: Reference formulation,1/2 tablet PO in fasted state D: 20 mg LY3337641 (T2fasted),1 tablet PO in fasted state B: 20 mg LY3337641 (T1fasted), 1 tablet PO in fasted state C: 20 mg LY3337641 (T1fed),1 tablet PO in fed state
- Sequence BACD: B: 20 mg LY3337641 (T1fasted), 1 tablet PO in fasted state A: Reference formulation,1/2 tablet PO in fasted state C: 20 mg LY3337641 (T1fed),1 tablet PO in fed state D: 20 mg LY3337641 (T2fasted),1 tablet PO in fasted state
- Sequence CBDA: C: 20 mg LY3337641 (T1fed),1 tablet PO in fed state B: 20 mg LY3337641 (T1fasted), 1 tablet PO in fasted state D: 20 mg LY3337641 (T2fasted),1 tablet PO in fasted state A: Reference formulation,1/2 tablet PO in fasted state
- Sequence DCAB: D: 20 mg LY3337641(T2fasted),1 tablet PO in fasted state C: 20 mg LY3337641 (T1fed),1 tablet PO in fed state A: Reference formulation,1/2 tablet PO in fasted state B: 20 mg LY3337641 (T1fasted), 1 tablet PO in fasted state
Period: Period 1
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 7 | 7 | 8
Received at Least 1 Dose of Study Drug | 7 | 7 | 7 | 8
Completed | 7 | 7 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 7 | 7 | 8
Completed | 7 | 6 | 7 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — scheduling conflict | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 6 | 7 | 8
Completed | 7 | 6 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 6 | 7 | 8
Completed | 7 | 5 | 7 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 5 | 7 | 8
Completed | 7 | 5 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Wash-out
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 5 | 7 | 8
Completed | 7 | 5 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence ADBC | Sequence BACD | Sequence CBDA | Sequence DCAB
Started | 7 | 5 | 7 | 8
Completed | 7 | 5 | 7 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Overall
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 29
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 25.53 (2.69)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3337641
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3337641
Time Frame: Period 1,2,3,4 (Day 1): Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48 and 72 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Reference Formulation (R-fasted): A single, PO dose reference formulation (R) with water after an overnight fast in one of four periods.
- LY3337641 (T1-fasted): A single, PO dose of 20 mg LY3337641 (T1) with water after an overnight fast in one of four periods.
- LY3337641 (T1-fed): A single, PO dose of 20 mg LY3337641 (T1) with water after a high fat meal in one of four periods.
- LY3337641 (T2-fasted): A single, PO dose of 20 mg LY3337641 (T2)with water after an overnight fast in one of four periods.
Arm/Group | Reference Formulation (R-fasted) | LY3337641 (T1-fasted) | LY3337641 (T1-fed) | LY3337641 (T2-fasted)
Number analyzed (Participants) | 28 | 29 | 27 | 27
nanograms per milliliter (ng/mL) | 66.7 (40) | 64.9 (41) | 56.8 (44) | 65.5 (35)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3337641
Description: Pharmacokinetics (PK): Area Under the Concentration versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of LY3337641
Time Frame: Period 1,2,3,4 (Day 1): Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48 and 72 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Reference Formulation (R-fasted) | LY3337641 (T1-fasted) | LY3337641 (T1-fed) | LY3337641 (T2-fasted)
Number analyzed (Participants) | 28 | 29 | 27 | 27
nanograms*hour per milliliter (ng*h/mL) | 373 (44) | 371 (47) | 351 (42) | 361 (43)

ADVERSE EVENTS:
Time Frame: 2 months
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Reference Formulation (R-fasted) | LY3337641 (T1-fasted) | LY3337641 (T1-fed) | LY3337641 (T2-fasted)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 6/28 | 4/29 | 5/27 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Formulation (R-fasted) (N=28) | LY3337641 (T1-fasted) (N=29) | LY3337641 (T1-fed) (N=27) | LY3337641 (T2-fasted) (N=27)
Catheter site bruise (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Catheter site swelling (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT03099148/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03099148/SAP_001.pdf